CLINICAL TRIAL: NCT00439205
Title: Oral Tumor Margin Detection Using Optical Spectroscopy
Brief Title: Oral Margin Spectroscopy Detection Using Optical Spectroscopy
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2006-0673; 1R21DE016485-01 (NIH)
Record Dates: First submitted 2007-02-21; First posted 2007-02-23 (Estimated); Last update posted 2017-10-20 (Actual); Status verified 2017-10

CONDITIONS: Oral Tumors
Keywords: Oral Tumors; Oral Margin Spectroscopy; Oral Spectroscopy; Optical Spectroscopy; Oral neoplastic lesions; FastEEM4 System; Multispectral Digital Microscope; MDM; Nonstandard imaging technology

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue removal and study biopsies to be done so that researchers can better compare the appearance and diagnosis at these sites to the images that were taken.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- MDM + FastEEM4: Multispectral digital microscope (MDM) + FastEEM4 Systems
  Interventions: Device: FastEEM4 System; Device: Multispectral Digital Microscope

INTERVENTIONS:
Device: FastEEM4 System — The FastEEM4 probe is moved toward the edge of the lesion(s) until it measures what appears to be normal mouth tissue.
Device: Multispectral Digital Microscope — The MDM instrument will take pictures of abnormal-appearing and normal-appearing areas in the mouth.
  Other Names: MDM

SUMMARY:
The goal of this clinical research study is to evaluate an imaging technology that may help clinicians see how far an area of pre-cancerous or cancerous tissue extends in the mouth.

DETAILED DESCRIPTION:
Fluorescence and Reflectance:

All tissue and cells are made up of tiny particles that give off small amounts of light. This light is called fluorescence. Cancerous cells and normal cells give off different amounts and types of fluorescence and also reflect (bounce back) light differently. Researchers want to better understand if fluorescence and reflectance from mouth tissue can be used to tell which cells are abnormal. This information may help doctors detect early mouth cancers and treat all areas affected by cancerous changes.

The MDM Instrument, FastEEM4 Instrument, POS Instrument, PS2 Instrument, and the IMS Instrument:

Five (5) instruments have been developed:

* the multispectral digital microscope (MDM), a microscope that allows fluorescence and reflectance to be collected;
* the FastEEM4, which can shine different colors of light on the mucosa (the lining of the mouth), which allows fluorescence and reflectance to be collected and looked at without surgically removing any tissue;
* the portable optical spectroscopy (POS) instrument, which is a smaller, portable version of the FastEEM4 device;
* the portable screening system (PS2), which can take images and measurements both in reflectance and in fluorescence mode; and
* the image mapping spectrometer (IMS), which is PS2 and POS combined.

The MDM system is a modified standard medical microscope similar to what doctors use to examine people's ears. A special light source has been attached to this microscope to provide different colors of light that can shine in the mouth. This microscope also has a digital camera attached to it so that researchers can take pictures of fluorescence and reflectance in the mouth in order to record what is seen with the different light colors. Researchers want to study the pictures in order to better understand the differences in fluorescence and reflectance from normal and abnormal cells.

The PS2 is an imaging device for examining the mouth without touching the mouth. The PS2 uses a blue light source in fluorescence mode. The light passes through a filter and shines on the tissue area. A filter is placed in the path to collect only the fluorescent light given off from the tissue. In reflectance mode, a white light is used. Images are collected using a device and a laptop with a software interface. A set of fluorescence and reflectance images can be taken in less than a minute.

The IMS is also an imaging device for examining the mouth without touching the mouth. The IMS includes white and blue light, a camera lens, customized optics (mirror, prisms, and lenses), a filter, a camera, and a computer. In reflectance mode, a white light shines on the tissue area, and specialized optics put the data on the camera. In fluorescence mode, the blue light highlights the tissue. A filter blocks the blue light, which allows tissue fluorescence to be seen. The IMS uses the same light sources as the PS2.

The FastEEM4 system (nonstandard imaging technology) has a probe (a small device used for measuring and/or detecting) that is about the size of a pencil. The probe is placed gently against the mucosa, and different colors of light are directed through the probe to a small area (the lesion and the normal-appearing area) of mouth tissue. Then the fluorescence and reflectance is recorded by a computer.

The POS instrument will direct different colors of light through fibers to the lining of the mouth and then light is collected and sent to a special camera and a computer to be analyzed. The spectroscopy system has a small probe about the size of a writing pen which is placed gently against the lining of the mouth. The exposed tissues will give off very small amounts of fluorescence. This light cannot be seen by the eye, but is seen by a computer.

Use of the MDM, PS2, or IMS Instruments:

If you agree to take part in this study, a clinician may first use the MDM, PS2, or IMSsystem. If one of these systems are used, the clinician will examine the inside of your mouth with a gloved finger while using standard white light or one or more of the imaging systems for viewing. The instrument will then take pictures of abnormal-appearing and normal-appearing areas in the mouth. The edge between these areas will then be marked with a surgical pen to outline the border between the abnormal-appearing tissue and normal-appearing tissue to be seen on a digital photo. Imaging with each device will take about 2 minutes or less. Between each use of the instrument, it will be sterilized according to standard practices.

Use of the FastEEM4 and/or POS Instruments:

The clinician may then use the FastEEM4 and/or the POS systems. If the FastEEM4 and/or POS systems are used, you will have a FastEEM4 and/or POS probe(s) placed gently on the mouth lesion(s). Several measurements will then be taken by moving the probe(s) a short distance at a time, toward the edge of the lesion(s), until it measures what appears to be normal mouth tissue.

Biopsies and Tissue Removal:

You may be having surgery to remove abnormal-appearing mouth lesions as part of standard care, so the study biopsies and tissue removal may be done at the same time as your surgery. After the surgeon has finished surgery and removed tissue from your mouth as part of your standard treatment, a portion of tissue (from both the abnormal-appearing and normal-appearing areas) that was already removed by the surgeon may be separated out from the main tissue specimen and separately evaluated. This is done so that the researchers can better compare the appearance and diagnosis at these sites to the images that were taken. In addition, a biopsy may be taken from the area of normal-appearing tissue from the opposite side of the mouth that was imaged with the FastEEM4 and/or POS probe(s), if the FastEEM4 and/or POS system(s) were used. If it is performed, this one biopsy of normal appearing tissue will be in addition to what is removed for standard care.

If this biopsy is performed, a small sample (4 mm, about the size of a small pencil eraser) of the lining of your mouth will be removed, while you are asleep under general anesthesia, from the area of normal-appearing tissue from the opposite side of the mouth that was imaged by both instruments.

Length of Study:

You will not be told of any experimental findings of this study. Information about the diagnosis will be available to your treating doctor. After tissue collection is complete, your participation in this study will be over.

All data (such as the tissue images and pathologic diagnosis) will be coded with a number instead of your personal identifying information (such as your name or medical record number) to help ensure your privacy.

This is an investigational study. Up to 60 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a lesion or history of a lesion of the oral mucosa.
2. Subjects with the ability and willingness to sign an informed consent and authorization.

Exclusion Criteria:

1. Persons who are medically unfit to undergo surgery.
2. Persons under the age of 18.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with precancerous or cancerous oral lesions.
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2007-02-07 (Actual); Primary Completion 2017-10-10 (Actual); Study Completion 2017-10-10 (Actual)

PRIMARY OUTCOMES:
Feasibility of using optical imaging and spectroscopy to assist in margin detection for tumor resection in the oral cavity. | 3 Years

CONTACTS AND LOCATIONS:
Overall Officials: Ann M. Gillenwater, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org